CLINICAL TRIAL: NCT05671497
Title: Evaluation of the Effect of Cilostazol on the Clinical Outcomes of Rheumatoid Arthritis Patients
Brief Title: The Effect of Cilostazol on Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other); Al-Azhar University (Other)
Responsible Party: Principal Investigator, Omar Ashraf Mohamed, Teaching Assistant, Misr International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACUC-FP-ASU
Record Dates: First submitted 2022-12-14; First posted 2023-01-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Cilostazol
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol arm (Experimental): 35 patients receiving conventional synthetic disease modifying antirheumatic drugs in addition to Cilostazol 100 mg twice daily for 6 months.
  Interventions: Drug: Cilostazol 100 MG; Drug: conventional synthetic antirheumatic drugs
- Control (Active Comparator): 35 patients receiving conventional synthetic disease modifying antirheumatic drugs for 6 months.
  Interventions: Drug: conventional synthetic antirheumatic drugs

INTERVENTIONS:
Drug: Cilostazol 100 MG — An antiplatelet agent used for intermittent claudication , it has an anti-inflammatory effect which will help control patients with Rheumatoid arthritis
  Arms: Cilostazol arm
Drug: conventional synthetic antirheumatic drugs — methotrexate 7.5-15 mg once weekly hydroxychloroquine 200 mg twice daily sulfasalazine 500 mg to 3 g once daily leflunomide 20 mg once daily

SUMMARY:
The goal of this study is to evaluate the effect of cilostazol on Rheumatoid Arthritis patients. It aims to answer the questions of :

1. Will Cilostazol improve the disease severity and quality of life in Rheumatoid arthritis patients?
2. Will Cilostazol decrease the oxidative stress, inflammation and endothelial dysfunction in Rheumatoid arthritis patients?

Participants will be randomized into two arms either treatment or control the treatment group will be asked to take Cilostazol 100 mg twice daily in addition to the usual DMARD (Methotrexate , Sulfasalazine , Hydroxychloroquine or Leflunomide), while the control group will be taking the usual DMARDs only.

Patients in both arms will be followed-up every 2 weeks through out the 6-month duration of the study.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is an autoimmune disease affecting joints. It usually affects females more. The available treatment aims to slow down disease progression and control the disease symptoms. Treatment is classified into either the conventional DMARDs (Methotrexate , Sulfasalazine , Hydroxychloroquine or Leflunomide) or Biological DMARDs such as an Anti-TNF alpha ( Certolizumab, Infliximab , Etanercept or Golimumab) or non-TNF biologics (Rituximab, Abatacept or Tocilizumab). Both classes have their drawbacks. The conventional DMARDs is not effective for many patients and the biological DMARDs have a high cost making their use limited to patients with medical insurance or patients who can afford it, thus making it necessary to find new medications which can improve the outcomes in patients with RA.

Cilostazol is an antiplatelet agent used mainly for intermittent Claudication. Recently many preclinical trials have shown efficacy of cilostazol in RA via it's anti-inflammatory action. it also decreases the oxidative stress which is high in ٌRA patients.

Patients will be randomized into two arms , one which is treatment and the other is control the treatment group will be asked to take Cilostazol 100 mg twice daily in addition to the usual DMARD (Methotrexate , Sulfasalazine , Hydroxychloroquine or Leflunomide), while the control group will be taking the usual DMARDs only.

Patients in both arms will be followed-up every 2 weeks through out the 6-month duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients. (>18 years old).
2. Moderate to high disease activity (DAS28-CRP>3.2).
3. Patients receiving stable cDMARD regimen for at least 3 months before inclusion in the study.

Exclusion Criteria:

1. Hypersensitivity to cilostazol.
2. Heart failure.
3. Pregnant and lactating women.
4. Patients with liver impairment (ALT or AST > 3* ULN).
5. Patients with renal impairment (CrCl<60 mL/min).
6. Patients receiving any other antiplatelet or anticoagulant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in the DAS-28 CRP score | Baseline, after 3 months , After 6 months
  DAS-28 score is used to asses disease severity in Rheumatoid Arthritis. It incorporates the swollen and tender joints present in 28 joints together with the c-reactive protein measurement into an equation to calculate the disease severity.
  0.56*
  √(TJC28) + 0.28* √(SJC28) + 0.36*ln (CRP + 1) +0.014*(GH) + 0.96
  where TJC:is tender joint count SJC is : swollen joint count GH:patient assessment of disease activity using a 100 mm visual analogue scale (VAS) with 0 = best, 100 = worst
  a number is given which is equal to a specific disease severity.
  website to calculate the DAS-28 score : https://www.4s-dawn.com/DAS28/

SECONDARY OUTCOMES:
Health Assessment Questionnaire | Baseline, after 3 months , After 6 months
  Rheumatoid arthritis health assessment questionnaire is a self-administered questionnaire help assess patients' functional status. Health assessment questionnaire is validated and present in Arabic language to be administered to Egyptian patients.
  There are 8 categories in the HAQ assessing the daily activities. In each category the highest score is taken. There are 2 to 3 questions in each category with a scale from 0 to 3 where 0 means no functional limitation and 3 means unable to do this activity. If the patient is using an assistive device the minimum score for this category should be 2. At the end the patient category score is added and divided by 8. The final score is given from 0 to 3 where 3 indicates a poor quality of life.
Total antioxidant capacity (TAC) | Baseline and at 6 months
  Oxidative stress is linked to the pathogenesis of various diseases including RA, cilostazol was shown to decrease the oxidative stress in other disease. so measuring the total antioxidant capacity in order to show the oxidative stress levels.
Malondialdehyde (MDA) | Baseline and at 6 months
  Malondialdehyde is a reactive oxygen species molecule. the level of MDA reflect the oxidative stress present which is important for the pathogenesis of various diseases including Rheumatoid arthritis
TNF α | Baseline and at 6 months
  TNF-alpha is a pro-inflammatory marker used to detect degree of inflammation , and as Rheumatoid arthritis is an inflammatory disease , TNF-alpha measurement would give an insight to RA inflammatory state. TNF-alpha is
phosphorylated Adenosine monophosphate-activated protein kinase (p-AMPK) | Baseline and at 6 months
  p-AMPK is an important marker of inflammatory response as it inhibits inflammatory pathway, measuring p-AMPK would give an insight on the inflammatory response present in Rheumatoid arthritis
Vascular cell adhesion protein 1(VCAM-1) | baseline and at 6 months
  ilostazol was reported to improve the endothelial dysfunction associated with diabetes in diabetic rats through decreasing the adhesion molecules, such as VCAM-1 by an AMPK dependent action which could be beneficial in RA associated endothelial dysfunction
Cilostazol safety | From date of randomization then every two weeks up to 6 months
  Cilostazol safety will be monitored by asking patients through monthly visits and using phone calls every 2 weeks about occurrence of any side effects. The expected side effects of cilostazol are; headache, diarrhea and nausea and stomach pain. Some serious side effects can occur such as bruising , bleeding , palpations and swelling of the arms, hands, feet, ankles, or lower legs

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahraa Hospital, Cairo, Egypt

REFERENCES:
- [Background] Almutairi K, Nossent J, Preen D, Keen H, Inderjeeth C. The global prevalence of rheumatoid arthritis: a meta-analysis based on a systematic review. Rheumatol Int. 2021 May;41(5):863-877. doi: 10.1007/s00296-020-04731-0. Epub 2020 Nov 11. PMID 33175207
- [Background] Castrejon I, Ortiz AM, Toledano E, Castaneda S, Garcia-Vadillo A, Patino E, Gonzalez-Alvaro I. Estimated cutoff points for the 28-joint disease activity score based on C-reactive protein in a longitudinal register of early arthritis. J Rheumatol. 2010 Jul;37(7):1439-43. doi: 10.3899/jrheum.091333. Epub 2010 May 15. PMID 20472931
- [Background] Cha Y, Erez T, Reynolds IJ, Kumar D, Ross J, Koytiger G, Kusko R, Zeskind B, Risso S, Kagan E, Papapetropoulos S, Grossman I, Laifenfeld D. Drug repurposing from the perspective of pharmaceutical companies. Br J Pharmacol. 2018 Jan;175(2):168-180. doi: 10.1111/bph.13798. Epub 2017 May 18. PMID 28369768
- [Background] Conigliaro P, Triggianese P, De Martino E, Fonti GL, Chimenti MS, Sunzini F, Viola A, Canofari C, Perricone R. Challenges in the treatment of Rheumatoid Arthritis. Autoimmun Rev. 2019 Jul;18(7):706-713. doi: 10.1016/j.autrev.2019.05.007. Epub 2019 May 3. PMID 31059844
- [Background] da Motta NA, de Brito FC. Cilostazol exerts antiplatelet and anti-inflammatory effects through AMPK activation and NF-kB inhibition on hypercholesterolemic rats. Fundam Clin Pharmacol. 2016 Aug;30(4):327-37. doi: 10.1111/fcp.12195. Epub 2016 Mar 31. PMID 26950185
- [Background] Das DC, Jahan I, Uddin MG, Hossain MM, Chowdhury MAZ, Fardous Z, Rahman MM, Kabir AKMH, Deb SR, Siddique MAB, Das A. Serum CRP, MDA, Vitamin C, and Trace Elements in Bangladeshi Patients with Rheumatoid Arthritis. Biol Trace Elem Res. 2021 Jan;199(1):76-84. doi: 10.1007/s12011-020-02142-7. Epub 2020 Apr 18. PMID 32306287
- [Background] Ferro F, Elefante E, Luciano N, Talarico R, Todoerti M. One year in review 2017: novelties in the treatment of rheumatoid arthritis. Clin Exp Rheumatol. 2017 Sep-Oct;35(5):721-734. Epub 2017 Sep 13. PMID 28956527
- [Background] Foster W, Carruthers D, Lip GY, Blann AD. Inflammatory cytokines, endothelial markers and adhesion molecules in rheumatoid arthritis: effect of intensive anti-inflammatory treatment. J Thromb Thrombolysis. 2010 May;29(4):437-42. doi: 10.1007/s11239-009-0370-y. PMID 19578810
- [Background] Fries JF, Spitz P, Kraines RG, Holman HR. Measurement of patient outcome in arthritis. Arthritis Rheum. 1980 Feb;23(2):137-45. doi: 10.1002/art.1780230202. PMID 7362664
- [Background] Gaffo A, Saag KG, Curtis JR. Treatment of rheumatoid arthritis. Am J Health Syst Pharm. 2006 Dec 15;63(24):2451-65. doi: 10.2146/ajhp050514. PMID 17158693
- [Background] Garcia-Gonzalez A, Gaxiola-Robles R, Zenteno-Savin T. Oxidative stress in patients with rheumatoid arthritis. Rev Invest Clin. 2015 Jan-Feb;67(1):46-53. PMID 25857584
- [Background] Kim HY, Lee SW, Park SY, Baek SH, Lee CW, Hong KW, Kim CD. Efficacy of concurrent administration of cilostazol and methotrexate in rheumatoid arthritis: pharmacologic and clinical significance. Life Sci. 2012 Sep 17;91(7-8):250-7. doi: 10.1016/j.lfs.2012.07.003. Epub 2012 Jul 20. PMID 22820172
- [Background] Lee YS, Lee SY, Park SY, Lee SW, Hong KW, Kim CD. Cilostazol add-on therapy for celecoxib synergistically inhibits proinflammatory cytokines by activating IL-10 and SOCS3 in the synovial fibroblasts of patients with rheumatoid arthritis. Inflammopharmacology. 2019 Dec;27(6):1205-1216. doi: 10.1007/s10787-019-00605-5. Epub 2019 May 23. PMID 31123968
- [Background] Lin YJ, Anzaghe M, Schulke S. Update on the Pathomechanism, Diagnosis, and Treatment Options for Rheumatoid Arthritis. Cells. 2020 Apr 3;9(4):880. doi: 10.3390/cells9040880. PMID 32260219
- [Background] Liu T, Zhang L, Joo D, Sun SC. NF-kappaB signaling in inflammation. Signal Transduct Target Ther. 2017;2:17023-. doi: 10.1038/sigtrans.2017.23. Epub 2017 Jul 14. PMID 29158945
- [Background] Matcham F, Scott IC, Rayner L, Hotopf M, Kingsley GH, Norton S, Scott DL, Steer S. The impact of rheumatoid arthritis on quality-of-life assessed using the SF-36: a systematic review and meta-analysis. Semin Arthritis Rheum. 2014 Oct;44(2):123-30. doi: 10.1016/j.semarthrit.2014.05.001. Epub 2014 May 29. PMID 24973898
- [Background] El Meidany YM, El Gaafary MM, Ahmed I. Cross-cultural adaptation and validation of an Arabic Health Assessment Questionnaire for use in rheumatoid arthritis patients. Joint Bone Spine. 2003 Jun;70(3):195-202. doi: 10.1016/s1297-319x(03)00004-6. PMID 12814762
- [Background] Noack M, Miossec P. Selected cytokine pathways in rheumatoid arthritis. Semin Immunopathol. 2017 Jun;39(4):365-383. doi: 10.1007/s00281-017-0619-z. Epub 2017 Feb 17. PMID 28213794
- [Background] Picerno V, Ferro F, Adinolfi A, Valentini E, Tani C, Alunno A. One year in review: the pathogenesis of rheumatoid arthritis. Clin Exp Rheumatol. 2015 Jul-Aug;33(4):551-8. Epub 2015 Jul 21. PMID 26203933
- [Background] Pisetsky DS. Advances in the Treatment of Rheumatoid Arthritis: Costs and Challenges. N C Med J. 2017 Sep-Oct;78(5):337-340. doi: 10.18043/ncm.78.5.337. PMID 28963273
- [Background] Pushpakom S, Iorio F, Eyers PA, Escott KJ, Hopper S, Wells A, Doig A, Guilliams T, Latimer J, McNamee C, Norris A, Sanseau P, Cavalla D, Pirmohamed M. Drug repurposing: progress, challenges and recommendations. Nat Rev Drug Discov. 2019 Jan;18(1):41-58. doi: 10.1038/nrd.2018.168. Epub 2018 Oct 12. PMID 30310233
- [Background] Refaie MMM, Ahmed Ibrahim R, Shehata S. Dose dependent effect of cilostazol in induced testicular ischemia reperfusion via modulation of HIF/VEGF and cAMP/SIRT1 pathways. Int Immunopharmacol. 2021 Dec;101(Pt A):108197. doi: 10.1016/j.intimp.2021.108197. Epub 2021 Oct 6. PMID 34626874
- [Background] Salminen A, Hyttinen JM, Kaarniranta K. AMP-activated protein kinase inhibits NF-kappaB signaling and inflammation: impact on healthspan and lifespan. J Mol Med (Berl). 2011 Jul;89(7):667-76. doi: 10.1007/s00109-011-0748-0. Epub 2011 Mar 23. PMID 21431325
- [Background] Samimi Z, Kardideh B, Zafari P, Bahrehmand F, Roghani SA, Taghadosi M. The impaired gene expression of adenosine monophosphate-activated kinase (AMPK), a key metabolic enzyme in leukocytes of newly diagnosed rheumatoid arthritis patients. Mol Biol Rep. 2019 Dec;46(6):6353-6360. doi: 10.1007/s11033-019-05078-x. Epub 2019 Nov 18. PMID 31541390
- [Background] Sarban S, Kocyigit A, Yazar M, Isikan UE. Plasma total antioxidant capacity, lipid peroxidation, and erythrocyte antioxidant enzyme activities in patients with rheumatoid arthritis and osteoarthritis. Clin Biochem. 2005 Nov;38(11):981-6. doi: 10.1016/j.clinbiochem.2005.08.003. Epub 2005 Sep 16. PMID 16150434
- [Background] Sorkin EM, Markham A. Cilostazol. Drugs Aging. 1999 Jan;14(1):63-71; discussion 72-3. doi: 10.2165/00002512-199914010-00005. PMID 10069409
- [Background] Sparks JA. Rheumatoid Arthritis. Ann Intern Med. 2019 Jan 1;170(1):ITC1-ITC16. doi: 10.7326/AITC201901010. PMID 30596879
- [Background] Suzuki K, Uchida K, Nakanishi N, Hattori Y. Cilostazol activates AMP-activated protein kinase and restores endothelial function in diabetes. Am J Hypertens. 2008 Apr;21(4):451-7. doi: 10.1038/ajh.2008.6. Epub 2008 Feb 7. PMID 18369362
- [Background] Usenbo A, Kramer V, Young T, Musekiwa A. Prevalence of Arthritis in Africa: A Systematic Review and Meta-Analysis. PLoS One. 2015 Aug 4;10(8):e0133858. doi: 10.1371/journal.pone.0133858. eCollection 2015. PMID 26241756
- [Background] van Gestel AM, Haagsma CJ, van Riel PL. Validation of rheumatoid arthritis improvement criteria that include simplified joint counts. Arthritis Rheum. 1998 Oct;41(10):1845-50. doi: 10.1002/1529-0131(199810)41:103.0.CO;2-K. PMID 9778226
- [Background] Charles J, Britt H, Pan Y. Rheumatoid arthritis. Aust Fam Physician. 2013 Nov;42(11):765. PMID 24217093
- [Background] Yoshida Y, Tanaka T. Interleukin 6 and rheumatoid arthritis. Biomed Res Int. 2014;2014:698313. doi: 10.1155/2014/698313. Epub 2014 Jan 12. PMID 24524085